CLINICAL TRIAL: NCT00548444
Title: Measurement of Human T-Cell Turnover Following Vaccination With the Tuberculosis Vaccine MVA85A
Brief Title: T-Cell Turnover Following Vaccination With MVA85A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); St George's, University of London (Other)
Responsible Party: Ms. Heather House, Head, Clinical Trials and Research Governance Office, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB018; EudraCT number: 2007-001293-8
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Lymphocyte kinetics; MVA85A; Deuterium
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Volunteers will receive a single dose of MVA85A followed by regular blood tests to measure the resulting cellular immune response.
  Interventions: Biological: MVA85A
- Group 2 (Experimental): Volunteers will receive a single dose of MVA85A followed by an infusion of labelled (deuterated) glucose and regular blood tests.
  Interventions: Biological: MVA85A; Other: Deuterated glucose infusion
- Group 3 (Experimental): Volunteers will receive a single dose of MVA85A followed by an infusion of labelled (deuterated) glucose and regular blood tests.
  Interventions: Biological: MVA85A; Other: Deuterated glucose infusion

INTERVENTIONS:
Biological: MVA85A — Vaccine. Dose: 1 x 10^8 plaque-forming units (pfu) given by intradermal injection into the deltoid region of the upper arm.
Other: Deuterated glucose infusion — 6,6D2-glucose given as a timed intravenous infusion. The total dose of deuterated glucose will be 1g/kg volunteer body weight (up to a maximum of 60g).
  Arms: Group 2; Group 3

SUMMARY:
This study examines the early immune response to a new vaccine (MVA85A) being developed to combat tuberculosis (TB).

DETAILED DESCRIPTION:
MVA85A is a promising new vaccine designed to prevent tuberculosis (TB) by dramatically boosting pre-existing responses to BCG, the only licensed vaccine against the disease at present. In BCG vaccinated individuals it induces a strong immune response. However little is known about the evolution of that response or of the kinetics of T-cells (the immune cells that respond to the vaccine) immediately following vaccination. Crucially, the outcome of this process may determine long term protection from disease.

This study aims to define the early immune response to MVA85A and is the first to apply a safe, non-radioactive 'label' - deuterium - to measure T-cell turnover following vaccination. This labelling approach has been used successfully by the study collaborators to examine immune cell kinetics in human clinical studies in the UK over the last 8 years. The resulting data will provide insight into the immune response generated by MVA85A and aid in the future design and modification of other T-cell inducing vaccines.

Group 1 (Immune responses only)

Previous human studies of MVA85A have described the immune response to vaccination at fixed timepoints but not in between. The investigators will vaccinate four volunteers and measure immune responses daily for 14 days. This will provide important new data and aid interpretation of kinetics data from groups 2 and 3.

Groups 2 & 3 (Labelling)

Eight volunteers will be vaccinated and then receive a timed infusion of deuterated glucose. Blood will be collected during the follow up period to determine the rates of uptake and loss of label in responding immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 50 years
* Immunization with BCG greater than 12 months prior to enrolment in the study
* Resident in or near Oxford for the duration of the study
* Able and willing (in the investigator's opinion) to comply with all study requirements
* Given written informed consent
* Willing to allow the investigator to request medical information from, or discuss the volunteer's medical history with the volunteer's General Practitioner
* Willing to allow the investigator to register volunteer details with a confidential database to prevent concurrent entry into clinical trials
* For women only, willingness to practice continuous effective contraception during the study
* Agreement to refrain from blood donation during the course of the study

Exclusion Criteria:

Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period

* Prior receipt of a recombinant MVA vaccine
* Screening test suggesting the possibility of latent TB infection- i.e. Elispot positive (greater than 17 sfc/million PBMC) in any ESAT6 peptide or CFP10 peptide pool
* Any clinically significant abnormal finding on screening blood tests or urinalysis (see Appendix B for guidance on study reference ranges)
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Any history of anaphylaxis
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (antibodies to HCV)
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other chronic illness requiring hospital specialist supervision
* Any other significant disease, disorder or finding, which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate fully in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Proliferation and disappearance rates of responding antigen-specific T-cells | Within four weeks of vaccination

SECONDARY OUTCOMES:
Immunogenicity | Within three months of vaccination
Safety | Within three months of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Helen I McShane, MBBS, MRCP, BSc, PhD, Principal Investigator — University of Oxford; Adrian VS Hill, MA, BM BCh, DPhil, DM, Study Chair — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Macallan DC, Wallace D, Zhang Y, De Lara C, Worth AT, Ghattas H, Griffin GE, Beverley PC, Tough DF. Rapid turnover of effector-memory CD4(+) T cells in healthy humans. J Exp Med. 2004 Jul 19;200(2):255-60. doi: 10.1084/jem.20040341. Epub 2004 Jul 12. PMID 15249595
- [Background] Vukmanovic-Stejic M, Zhang Y, Cook JE, Fletcher JM, McQuaid A, Masters JE, Rustin MH, Taams LS, Beverley PC, Macallan DC, Akbar AN. Human CD4+ CD25hi Foxp3+ regulatory T cells are derived by rapid turnover of memory populations in vivo. J Clin Invest. 2006 Sep;116(9):2423-33. doi: 10.1172/JCI28941. PMID 16955142
- [Background] Asquith B, Zhang Y, Mosley AJ, de Lara CM, Wallace DL, Worth A, Kaftantzi L, Meekings K, Griffin GE, Tanaka Y, Tough DF, Beverley PC, Taylor GP, Macallan DC, Bangham CR. In vivo T lymphocyte dynamics in humans and the impact of human T-lymphotropic virus 1 infection. Proc Natl Acad Sci U S A. 2007 May 8;104(19):8035-40. doi: 10.1073/pnas.0608832104. Epub 2007 May 1. PMID 17483473
- [Background] McShane H, Pathan AA, Sander CR, Keating SM, Gilbert SC, Huygen K, Fletcher HA, Hill AV. Recombinant modified vaccinia virus Ankara expressing antigen 85A boosts BCG-primed and naturally acquired antimycobacterial immunity in humans. Nat Med. 2004 Nov;10(11):1240-4. doi: 10.1038/nm1128. Epub 2004 Oct 24. PMID 15502839